CLINICAL TRIAL: NCT01023698
Title: Panretinal Photocoagulation for Proliferative Diabetic Retinopathy in a Single Session Using Low Fluence Parameters
Acronym: PFC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC0003
Record Dates: First submitted 2009-11-26; First posted 2009-12-02 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Neovascular
Keywords: Diabetic retinopathy; Diabetic macular edema; Panretinal photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- photocoagulation (Experimental): Laser photocoagulation
  Interventions: Procedure: laser photocoagulation

INTERVENTIONS:
Procedure: laser photocoagulation — Laser photocoagulation

SUMMARY:
Is it possible to do a panretinal photocoagulation for proliferative diabetic retinopathy in a single session using low fluence parameters?

ELIGIBILITY:
Inclusion Criteria:

* untreated Proliferative diabetic retinopathy

Exclusion Criteria:

* Previous photocoagulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Stabilization of proliferative diabetic retinopathy | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Martinez-Castellanos, MD, Principal Investigator — Asociacion para Evitar la Ceguera en México